CLINICAL TRIAL: NCT06881056
Title: A Phase 2 Multicenter, Randomized, Open-label Study to Evaluate the Pharmacokinetic, Safety and Efficacy of Peginterferon Alfa-2b Injection in Subjects With Essential Thrombocythemia Who Are Resistant to or Intolerant of Hydroxyurea.
Brief Title: Peginterferon α-2b Injection for Aerosol Therapy in Pediatric Respiratory Syncytial Virus Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Lisa Moon, Chief physician, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y2024033
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Respiratory Syncytial Virus (RSV); Peginterferon α-2b injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peginterferon α-2b 45 mcg dose group (Experimental)
  Interventions: Drug: Peginterferon α-2b injection
- Peginterferon α-2b 90 mcg dose group (Experimental)
  Interventions: Drug: Peginterferon α-2b injection
- Control group (Other)
  Interventions: Behavioral: symptomatic and supportive treatment

INTERVENTIONS:
Drug: Peginterferon α-2b injection — Peginterferon α-2b injection, 45 mcg, neb.On the 1st, 3rd, and 5th day, take the medication,while providing symptomatic and supportive treatment simultaneously.
  Arms: Peginterferon α-2b 45 mcg dose group
Drug: Peginterferon α-2b injection — Peginterferon α-2b injection, 90 mcg, neb.On the 1st, 3rd, and 5th day, take the medication,while providing symptomatic and supportive treatment simultaneously.
  Arms: Peginterferon α-2b 90 mcg dose group
Behavioral: symptomatic and supportive treatment — symptomatic and supportive treatment
  Arms: Control group

SUMMARY:
This is a multicenter, randomized, open-label, parallel-controlled, prospective clinical study. It aims to evaluate the efficacy and safety of aerosolized Peginterferon α-2b injection in the treatment of pediatric respiratory syncytial virus pneumonia. The overall study is divided into a screening period, a treatment period, and a follow-up period. Eligible children with respiratory syncytial virus pneumonia will be randomly assigned to the experimental group 1, experimental group 2, and the control group at a ratio of 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age: 1 year ≤ age ≤ 3 years; (2) Gender: Both male and female participants are eligible; (3) According to the 9th edition of "Zhu Fute's Practical Pediatrics," meet the following diagnostic criteria: a. RSV test positive; b. Clinical manifestations: Fever, cough, wheezing; c. Physical signs: Rapid breathing and moist rales in the lungs; (4) Time: The time from the onset of the child's illness to the signing of the informed consent form is within 72 hours (starting from the occurrence of any symptom such as fever, cough, or wheezing); (5) Informed consent: The legal guardian of the child understands and signs the informed consent form (if the legal guardians are the parents, both parents need to sign together).

Exclusion Criteria:

* (1) Presence of any of the following clinical symptoms before enrollment: a. Poor general condition, with altered consciousness, refusal to eat, or signs of dehydration; b. Hypoxemia: Presence of cyanosis, rapid breathing (RR ≥ 50 breaths per minute), stridor, nasal flaring, tracheal tug, oxygen saturation < 92%, and intermittent apnea; c. Extrapulmonary complications; d. Chest X-ray or CT: Multilobar lung infiltrates, pleural effusion, pneumothorax, atelectasis, lung necrosis, and lung abscess; e. Hyperpyrexia: Persistent high fever for more than 5 days; f. Presence of critical complications such as respiratory failure and circulatory failure; (2) Allergy history and treatment history: a. Receiving antiviral drug treatment with interferon, ribavirin, acyclovir, ganciclovir, or vidarabine monophosphate within 30 days before screening or currently; b. Receiving immunoglobulin treatment within 30 days before screening or currently; c. Known hypersensitivity to interferon or its components, or a clear history of other allergies that make participation in this study inappropriate; d. Use of other investigational drugs within 3 months before screening or within 5 half-lives (whichever is longer), or currently participating in a clinical trial for a medical device at the time of screening; (3) Disease history and current medical history: a. History of congenital heart disease, severe malnutrition, abnormal immune system function, or other serious diseases of major organ systems; b. Severe liver or renal dysfunction; c. History of viral infections such as HBV, HCV, HIV; d. Past or current history of malignant tumors; e. Past history of epilepsy, or history and family history of neurological/psychiatric disorders; (4) Other conditions: Subjects deemed unsuitable for participation in this trial by the investigator.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time for the disappearance of major clinical symptoms | Day 6
  Major clinical symptoms include fever, cough, wheezing, increased respiratory rate, and moist rales in the lungs
The time of disappearance of abnormal signs. | Day 6
  Abnormal signs include fever, cough, wheezing, increased respiratory rate, and moist rales in the lungs.

SECONDARY OUTCOMES:
Compare the differences in treatment efficacy rates among the various groups. | Day 6
Compare the differences in the proportions of primary clinical symptoms alleviated/disappeared among the various groups. | Day3,5.
Compare the differences in the proportions of abnormal physical signs alleviated or disappeared among the various groups. | Day3,5.
Compare the differences in the time curves for the normalization of major clinical symptoms among the various groups. | Day6
Compare the differences in the time curves for the normalization of major abnormal physical signs among the various groups. | Day6
Compare the differences in total hospitalization duration among the various groups. | Day6

CONTACTS AND LOCATIONS:
Overall Officials: Lina Chen, Ph.D, Principal Investigator — West China Second University Hospital
Locations (2):
- China (2):
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - West China Second University Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No